CLINICAL TRIAL: NCT00646139
Title: A Combined Rising Single-Dose (RSD) and Rising Multiple-Dose (RMD) Phase 1 Study to Evaluate Safety, Tolerability and Pharmacokinetics of KX2-391 in Patients With Advanced Malignancies That Are Refractory to Conventional Therapies
Brief Title: KX2-391 in Treating Patients With Advanced Solid Tumors or Lymphoma That Did Not Respond to Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Alex Adjei, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000589972; RPCI-I-112607; KINEX-KX01-01-07
Record Dates: First submitted 2008-03-27; First posted 2008-03-28 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: Lymphoma; Lymphoproliferative Disorder; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; splenic marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; post-transplant lymphoproliferative disorder; cutaneous B-cell non-Hodgkin lymphoma; Waldenstrom macroglobulinemia; small intestine lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoproliferative Disorders; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Intraocular Lymphoma; Waldenstrom Macroglobulinemia | interventions — tirbanibulin; Immunoenzyme Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Src kinase inhibitor KX2-391
Other: immunoenzyme technique
Other: pharmacological study

SUMMARY:
RATIONALE: KX2-391 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of KX2-391 in treating patients with advanced solid tumors or lymphoma that did not respond to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To define the maximum tolerated dose of KX2-391 when administered as multiple oral solutions in patients with refractory advanced solid tumors and lymphoma.

Secondary

* To determine the safety and tolerability of KX2-391 given as single and multiple oral solutions in these patients.
* To characterize the pharmacokinetic profile of single dosing and multiple dosing of KX2-391 in these patients.
* To determine the biological effects of KX2-391.

OUTLINE: This is a multicenter study.

Patients receive oral KX2-391 once or twice daily for 3 weeks. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Blood and urine samples are collected periodically for pharmacokinetic studies. Biological effects are assessed by measuring plasma levels of vascular endothelial growth factor by ELISA. Levels of phospho-Src Tyr and transphosphorylation of selected substrates are measured in peripheral blood mononuclear cells.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of advanced solid tumor or lymphoma

  * Metastatic or unresectable disease
  * Standard curative or palliative measures do not exist or are no longer effective
* Patients with treated brain or ocular metastases are eligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 14 weeks
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Serum bilirubin ≤ 2.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Serum creatinine ≤ 1.5 times ULN or creatinine clearance > 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception for 1 month prior to, during, and for 6 months after completion of study treatment
* No inflammatory bowel disease, malabsorption syndrome, or other medical condition that may interfere with oral drug absorption
* No signs or symptoms of end organ failure, major chronic illnesses other than cancer, or any severe concomitant conditions including, but not limited to, active infections that, in the opinion of the investigator, precludes protocol participation or compliance
* No history of any of the following within the past 6 months:

  * Angina pectoris
  * Coronary artery disease
  * Hypertension
  * Cerebral vascular accident
  * Transient ischemic attack uncontrolled by medical therapy
* No history of confirmed cardiac conduction abnormalities or arrhythmias
* No known history of hepatitis B or C, or HIV infection
* No known history of coagulation disorders or hemolytic conditions (e.g., sickle cell anemia)

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* No prior major surgery to the upper gastrointestinal tract
* More than 2 weeks since prior investigational agents or systemic anticancer agents (28 days for agents with unknown elimination half-lives or known elimination half-lives > 50 hours)
* More than 4 weeks since prior radiotherapy to the sternum, pelvis, scapulae, vertebrae, or skull and recovered
* More than 4 weeks since prior major surgery
* More than 1 week since prior palliative low-dose radiotherapy to the limbs and recovered
* More than 2 weeks since prior and no concurrent hormones (e.g., estrogen contraceptives, hormone replacement, anti-estrogen, or progesterone) or antiplatelet agents
* More than 2 weeks since prior and no concurrent anticoagulants (e.g., coumadin) except prophylactic doses of anticoagulants for indwelling venous catheters
* More than 2 weeks or 5 half-lives since prior and no concurrent cytochrome P450 modulators (e.g., strong inducers or inhibitors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose

SECONDARY OUTCOMES:
Safety
Pharmacokinetics
Biological effects

CONTACTS AND LOCATIONS:
Overall Officials: Alex A. Adjei, MD, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States